CLINICAL TRIAL: NCT04251676
Title: Radiation Therapy in Uterine Cancer: Dosimetry Analysis, Clinical Implication, and Survival Analysis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201910019RINA
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study — Observational study

SUMMARY:
We wish to study radiation therapy in uterine cancer, focusing on dosimetry analysis, clinical implication, and survival analysis.

DETAILED DESCRIPTION:
We wish to study radiation therapy in uterine cancer, focusing on dosimetry analysis, clinical implication, and survival analysis.

ELIGIBILITY:
Inclusion Criteria:

* Women with uterine cancer (stage I - IV) treated in National Taiwan University Hospital, from January 2010 to September 2019.

Exclusion Criteria:

* Women with uterine cancer (stage I - IV) NOT treated in National Taiwan University Hospital, from January 2010 to September 2019.

Ages: 20 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women with uterine cancer (stage I - IV) treated in National Taiwan University Hospital, from January 2010 to September 2019.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 5 years
  Progression free survival: The time from inclusion to documented disease progression according to RECIST v1.1 or death from any cause.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen JL, Huang YS, Huang CY, Hsu CY, Lan KH, Cheng WF, Kuo SH. Impact of adjuvant radiotherapy on the survival of women with optimally resected stage III endometrial cancer in the era of modern radiotherapy: a retrospective study. Radiat Oncol. 2020 Apr 6;15(1):72. doi: 10.1186/s13014-020-01523-5. PMID 32252781